CLINICAL TRIAL: NCT07296549
Title: Expert Consensus on the Clinical Management of Melasma: A Delphi Method Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Melasma Consensus
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Melasma; Melasma (Facial Melasma)
Keywords: Melasma; consensus; expert panel; delphi method
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts participating in a Modified Delphi process to develop consensus recommendations on the management of melasma

SUMMARY:
This study aims to gather expert opinions on the best ways to treat and manage melasma, a common skin condition characterized by dark patches on the face. Using a method called the Delphi Method, a group of dermatologists and other specialists will participate in several rounds of surveys to share their insights and reach a consensus on the most effective treatments and management strategies. The goal is to create a set of evidence-based guidelines that can help doctors provide more consistent, effective care for patients with melasma. The study will ensure that all experts' opinions are anonymous, and the results will be shared to improve treatment practices worldwide.

DETAILED DESCRIPTION:
This study is designed to establish expert consensus on the management and treatment of melasma through a Delphi Method approach. The Delphi Method is a structured, iterative process where a panel of specialists-primarily dermatologists and other healthcare professionals experienced in treating melasma-will be asked to respond to a series of surveys. These surveys will allow experts to share their opinions on the most effective treatments, diagnostic criteria, and management strategies for melasma.

The study will be conducted in multiple rounds:

Round 1: Experts will provide open-ended feedback on their experiences and perspectives on melasma treatment.

Round 2: Based on the responses from Round 1, a refined set of questions will be circulated to clarify or expand on the issues raised.

Round 3: A final round will help refine and solidify the consensus on treatment approaches and care protocols.

The experts' feedback will be anonymized to ensure unbiased responses, and each round will be followed by analysis to identify areas of agreement and disagreement. The goal is to achieve a high level of consensus (usually around 70%) on key treatment recommendations and best practices for managing melasma.

This process will result in evidence-based guidelines for melasma treatment that healthcare providers can use to standardize care and improve patient outcomes. These guidelines will help address the variability in treatment practices and ensure that patients receive the most effective and up-to-date care based on expert consensus.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified or equivalent dermatologist,
* Minimum of 5 years of post-certification clinical experience in the management of MELASMA,
* Willingness to participate in all Delphi rounds.

Exclusion Criteria:

* Inability or unwillingness to complete Delphi rounds.
* Lack of clinical experience with MELASMA
* Industry representatives without direct clinical practice

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population:A purposive sample of experienced clinical dermatologists who actively manage melasma. The panel will include clinicians with diverse practice settings and geographic representation relevant to the study scope.Panel size and rationale:Target enrolment: 20-35 experts.Rationale: this size balances breadth of opinion and feasibility for iterative Delphi rounds; it is large enough to capture diverse viewpoints yet small enough to allow meaningful, anonymized feedback and analysis.Minimum required for analysis: 15 panelists
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Consensus on Diagnostic & therapeutic Criteria for Melasma | 6-12 weeks
  Establishment of expert consensus on core domains of melasma diagnosis and management measured by the proportion of statements reaching predefined consensus agreement after completion of delphi rounds

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged